CLINICAL TRIAL: NCT05302596
Title: Preserving Lean Body Mass During Weight Loss In Elderly Obese Patients With GLP-1 Receptor Agonist Treatment
Brief Title: Semaglutide Use in Elderly Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Husam A Ghanim, Research Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005760; UL1TR001412 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Aging
Keywords: Body composition; Adipose tissue; semaglutide
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, controlled, randomized and open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Semaglutide, added to standard of care, starting dose of 0.25mg titrated up to 1mg dose. for a total of 16 weeks.
  Interventions: Drug: Semaglutide Pen Injector
- standard of care only (No Intervention): Standard of Care (SOC) weight loss intervention alone (personalized lifestyle and exercise)

INTERVENTIONS:
Drug: Semaglutide Pen Injector — semaglutide (up to 1mg) once weekly injection added to the standard of care weight loss program. Semaglutide dose will be started at 0.25 mg dose during the baseline visit and doubled every 2 weeks up to 1mg dose or up to maximum tolerable dose for total of 16 weeks of intervention
  Other Names: Ozempic
  Arms: Semaglutide

SUMMARY:
This is a single-center, prospective, controlled, randomized and open label study to investigate the effect of the semaglutide addition to standard of care weight loss intervention (personalized lifestyle and exercise) in elderly obese subjects on body weight and body composition as assessed by DEXA.

DETAILED DESCRIPTION:
This will be a single center, prospective, open label, randomized and controlled pilot study to investigate the effects of semaglutide addition to a standard weight loss intervention program for 16 weeks on body weight and composition, adipose tissue metabolism and muscle strength compared to the standard weight loss program alone in elderly obese patients.

Eligible and qualified patients will be randomized 1:1 in pairs (8 pairs) matched by age and BMI within 5% and by gender to one of two open-label interventions. Priority of enrollment will be to match already existing and non-matched pair(s) before starting new ones. However, participants will not need to wait until they are matched to be enrolled in the study. The two open-label interventions are:

1. Control group: Standard of care weight loss program that includes lifestyle changes and personalized exercise and dietary education.
2. Semaglutide group: semaglutide (up to 1mg) once weekly injection added to the standard of care weight loss program. Semaglutide dose will be started at 0.25 mg dose during the baseline visit and doubled every 2 weeks up to 1mg dose or up to maximum tolerable dose. Patients will be instructed on how to inject themselves with the drug and how to increase the dose. During dose escalation, we will be monitoring the subject more extensively (4 weeks and 8 weeks), compared to clinical practice, for any side effects including if they experience any GI side effects, and subjects will be kept at the maximum tolerable dose up to 1mg/week.

At the baseline visit, and for all other visits, patients will come fasting (10 -12 hours) to the research center. Patients will visit the research center at 4 weeks (safety visit), 8 weeks and at 16 weeks (final study assessment visit). Blood (about 25 ml), body weight and other vitals, adverse events including hypoglycemia (blood sugar <70 mg/dl) will be collected at all visits. Fat biopsy aspiration, DEXA scans, muscle strength measurement and age-appropriate quality of life questionnaire (Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) will be performed at 0- and 16-weeks visits.

All patients will receive instructions at the beginning of the study on weight loss nutritional program and appropriate physical activity to be performed for the next 16 weeks. The program will be based, in-part, on dietary and exercise habits collected at screening visit. For the entire duration of the study, participants will maintain a daily diary to document food and exercise activities to ensure compliance with lifestyle program provided. At the 4- and 8-weeks visits, the daily diary will be reviewed for food and exercise activities, and instructions will be provided again to reinforce intervention.

Patients will be provided with glucose meter and glucose strips to measure fingerpick blood glucose. For the entire duration of the study, patients will be asked to measure their blood sugars at least one time after exercise and to record any hypoglycemic events (glucose <70mg/dl) in their diary, Patients will be instructed to record any other untoward side effects like nausea, vomiting, changes in appetite and other experiences in the diary. Patients will be instructed to call the Diabetes Center to speak to a study investigator directly in case of any problem or untoward side effects.

they have a question or side effects.

Standard of care weight loss program:

All patients will be instructed to implement dietary and exercise program for the next 16 weeks and to record their activities on daily food and exercise diary provided.

1. Energy intake should be reduced by 500-750kcal/day.
2. Dietary fat should be reduced to 30% of total energy intake maximally.
3. Meal replacements (if used) will be consumed during breakfast and lunch.
4. Dinner consisted of conventional food and participants will be encouraged to eat fruits and vegetables within their calorie limit.
5. Participants should ingest 1.0-1.5g of protein/kg/day and spread consumption equally throughout the day. A leucine-enriched balanced amino acid supplement can be used.
6. Subjects will be instructed to perform aerobic, muscle-strengthening, flexibility, and balance exercises. Minimally, this should include moderate-intensity aerobic activity for 30 minutes five days per week or vigorous-intensity aerobic activity for 20 minutes three days a week, 10-15 repetitions of 8-10 major muscle group strengthening exercises two or more nonconsecutive days each week, 10 minutes of flexibility activities at least two days a week, and balance exercises three times a week for fall prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age: ≥65 years
2. BMI ≥30 Kg/m2 AND waist circumference for women: > 80 cm and for men: > 90 cm
3. Stable body weight (no more than ±3 kg change during the 3 months prior to screening)
4. Able to participate in personalized physical activities and dietary instructions.
5. Participant must be able to read, write, and understand the English language and be able to provide written consent.

Exclusion Criteria:

1. Current diagnosis of weight changing condition including cancer, gastrointestinal conditions or eating disorders
2. GLP-1R agonists use within last 6 months
3. Diagnosis of type 1 or 2 diabetes
4. Impaired cognitive function (VA-St. Louis University Mental Survey (VA-SLUMS) score ≤ 19)
5. History of chronic/idiopathic acute pancreatitis
6. Personal/family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
7. Previous surgical treatment for obesity
8. Smoking or use of any nicotine products
9. Use of any medication that could interfere with trial results especially weight management drugs
10. Anticipated change in lifestyle (e.g., dietary, exercise or sleeping pattern) other than provided by the study.
11. Hepatic disease or cirrhosis
12. Aspartate Aminotransferase (AST) > 3X Upper limit of normal (ULN) and/or Alanine aminotransferase (ALT) > 3X ULN
13. Inability to give informed consent
14. History of gastroparesis
15. History of serious hypersensitivity reaction to these agents
16. Alcoholism
17. Patients with retinopathy
18. Participation in any other concurrent interventional clinical trial -

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Husam A Ghanim, PhD, Principal Investigator — State University of NY at Buffalo
Locations (1):
- Diabetes and Endocrinology Research Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semaglutide | Standard of Care Only
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Standard of Care Only | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (5.0) | 69.7 (5.1) | 69.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 38.2 (4.7) | 37.0 (4.3) | 37.8 (4.4)
Weight [Mean (Standard Deviation); unit: Kg] | 107.8 (19.8) | 100.0 (17.8) | 103.9 (19.5)
Total Fat Mass [Mean (Standard Deviation); unit: Kg] | 52.1 (8.9) | 47.8 (9.3) | 50.0 (9.0)
Total Fat-Free Mass [Mean (Standard Deviation); unit: Kg] | 51.0 (11.4) | 47.8 (6.4) | 49.4 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Body Composition as Total Fat Mass/ Total Fat-free Mass Ratio
Description: total fat mass/total fat-free mass ratio reported as arbitrary units (ratio), calculated by dividing total fat mass by total fat-free mass (lean mass) at baseline and at 16 weeks in both groups. Primary measurements of fat and fat-free mass is done using DEXA
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Arbitrary units (ratio)
Arm/Group | Semaglutide | Standard of Care Only
Number analyzed (Participants) | 7 | 7
Arbitrary units (ratio)
  Baseline | 1.04 (0.07) | 1.0 (0.07)
  16 Weeks | 0.96 (0.06) | 0.99 (0.07)

2. Primary Outcome: Body Weight
Description: body weight reported in Kg at at baseline and at 16 weeks in both groups
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Semaglutide | Standard of Care Only
Number analyzed (Participants) | 7 | 7
Kg
  Baseline | 107.8 (7.7) | 100.0 (6.7)
  16 weeks | 99.7 (7.2) | 97.1 (7.5)

3. Secondary Outcome: Total Fat Mass
Description: total fat mass reported in Kg and measured using DEXA at baseline and at 16 weeks in both groups
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Semaglutide | Standard of Care Only
Number analyzed (Participants) | 7 | 7
Kg
  Baseline | 52.1 (3.6) | 47.8 (3.9)
  16 weeks | 46.8 (3.6) | 46.3 (4.1)

4. Secondary Outcome: Total Fat-free Mass (Lean Mass)
Description: total fat-free mass (lean mass) reported in Kg and measured using DEXA at baseline and at 16 weeks in both groups
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Semaglutide | Standard of Care Only
Number analyzed (Participants) | 7 | 7
Kg
  baseline | 51.0 (4.2) | 47.8 (2.2)
  16 weeks | 49.5 (4.0) | 47.0 (2.4)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Semaglutide | Standard of Care Only
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 5/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=7) | Standard of Care Only (N=7)
Gastrointestinal side effects: constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) — constipation
GI side effects: Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) — Nausea
GI side effects: Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT05302596/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT05302596/ICF_001.pdf